CLINICAL TRIAL: NCT06426953
Title: Predictive Effect of TGF-β Combined With INS-PI3K-AKT Signaling Pathway Related Proteins (ADNP, MAP6, Pgc-1α) for POD in Diabetes Patients
Brief Title: Predictive Effect of TGF-β and INS-PI3K-AKT Related Proteins for POD in Diabetes Patients
Status: Recruiting | Type: Observational
Sponsor: Xie Kangjie (Other)
Responsible Party: Sponsor-Investigator, Xie Kangjie, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: IRB-2024-467（IIT）
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Postoperative Delirium
MeSH Terms: conditions — Diabetes Mellitus; Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A total of 3 mL peripheral blood samples were collected within 30 minutes before surgery and placed in a coagulation test tube at 4 °C. After centrifugation at 3000 rpm for 10 minutes at 4 °C, the plasma was separated, transferred into cryopreservation tubes, and stored at -80 °C. Upon collecting a sufficient number of samples, TGF-β, ADNP, MAP6, and PGC-1α were detected in the laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- History of diabetes ≥2 years and Glycated hemoglobin ≥6.5%: Diabetic patients with a history of more than 2 years
  Interventions: Other: No intervention
- No history of diabetes and normal blood glucose: Patients without a history of diabetes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To investigate the relationship between POD, TGF-β and INS-PI3K-AKT signaling pathway related proteins (ADNP, MAP6, PGC-1α) in diabetic patients

DETAILED DESCRIPTION:
The study was a two-center, prospective，single blind (blinded to subjects and evaluators)，control, observational clinical study. Participants will collect 3 milliliters of blood from enrolled patients before surgery begins. The collected blood samples were processed and stored in -80℃ refrigerator. All samples were tested TGF-β and INS-PI3K-AKT signaling pathway related proteins (ADNP, MAP6, PGC-1α) by ELISA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years
2. History of diabetes ≥2 years and Glycated hemoglobin ≥6.5% or no history of diabetes and normal blood glucose
3. The ASA rating is Class I to III
4. The elderly patients of limited thoracic and abdominal tumor surgery

Exclusion Criteria:

1. Refused to participate
2. Previous history of schizophrenia, epilepsy, Parkinson's disease
3. History of alcohol abuse or drug dependence
4. Patients with ASA grade IV and above
5. Severe visual or hearing impairment, can not cooperate with the completion of cognitive function tests
6. Participants in other clinical trials within the last two months
7. Patients with severe arrhythmia or cardiac dysfunction(EF<40%)
8. There was a clear history of neurological and psychiatric problems or long-term use of sedatives or antidepressants
9. History of cerebrovascular disease or brain surgery or trauma
10. Severe liver dysfunction (Child-Pugh class C) or severe renal dysfunction (requiring dialysis)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with a history of diabetes ≥2 years and a glycated hemoglobin of ≥6.5% or without a history of diabetes and a normal blood glucose level
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The correlation between preoperative plasma levels of TGF-β, ADNP, MAP6, PGC-1α and the incidence of delirium within 3 days after operation was analyzed. | 2024-05 to 2026-06
  Postoperative delirium (POD) was assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) and the 3-Minute Diagnostic Interview for Confusion Assessment Method-Defined Delirium (3D-CAM).
  Transforming growth factor-beta (TGF-β), activity-dependent neuroprotective protein (ADNP), microtubule-associated protein 6 (MAP6), and peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) levels were measured using enzyme-linked immunosorbent assay (ELISA) kits.

CONTACTS AND LOCATIONS:
Overall Officials: Kangjie Xie, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - The People's hospital of Qiannan, Duyun, Guizhou
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang